CLINICAL TRIAL: NCT01318161
Title: Epidural or Patient-controlled Analgesia for Colorectal Cancer Surgery. Long-term Outcomes.
Brief Title: Epidural Versus Patient-controlled Analgesia for Reduction in Long-term Mortality Following Colorectal Cancer Surgery
Acronym: EPICOL
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Difficulty in recruiting
Sponsor: Örebro University, Sweden (Other)
Collaborators: University Hospital, Linkoeping (Other)
Responsible Party: Principal Investigator, Anil Gupta, Associate Professor, Örebro University, Sweden
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2010/415-31
Record Dates: First submitted 2011-03-17; First posted 2011-03-18 (Estimated); Last update posted 2021-02-16 (Actual); Status verified 2021-02

CONDITIONS: Colorectal Cancer; Pain; Other Complications
Keywords: Epidural analgesia; Patient controlled analgesia; Colorectal cancer; Morbidity; Mortality
MeSH Terms: conditions — Colorectal Neoplasms; Pain | interventions — Ropivacaine; Morphine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Epidural anesthesia and analgesia (Experimental)
  Interventions: Drug: Ropivacaine + opioid epidurally
- Patient controlled analgesia (Active Comparator)
  Interventions: Drug: Morphine

INTERVENTIONS:
Drug: Ropivacaine + opioid epidurally — Epidural analgesia with local anesthetic + opioid
  Arms: Epidural anesthesia and analgesia
Drug: Morphine — Morphine via PCA pump
  Arms: Patient controlled analgesia

SUMMARY:
Colorectal cancer is one of the most common cancers in the industrialized world (12% of all cancers). In Sweden, 6000 new cases of colorectal cancer are reported each year, and almost half of these cases result in death. Several recently published retrospective studies show that regional anaesthesia (RA) can reduce cancer-related mortality following surgical treatment of colorectal, breast and prostate cancers and malignant melanoma. If these results are true, then the choice of perioperative pain management is as beneficial, or even better, than the current oncological therapies. This theory needs to be investigated in a prospective, randomized and controlled trail.

DETAILED DESCRIPTION:
An application was sent to the Regional Ethics Committee at the Linköping University Hospital and the study was approved recently. Informed consent will be obtained from 300 patients (ASA status 1-3) in the age group 40-80 years who are undergoing elective surgery for colorectal cancer. The exact type of cancer, its staging, degree of spread to proximal or distant sites and the pathologic type of cancer will be recorded. Patients on chronic narcotic analgesic medication, those with known immunologic diseases, those with known allergy to LA and those where epidural catheter placement is contraindicated will be excluded. This study will be a multi-centre study in Central Sweden. Patients will be randomized to one of two groups according to a computer-generated random number: Group E - Epidural anaesthesia (EDA) or Group P - Patient-controlled analgesia (PCA).

Anaesthesia and surgery will be standardized, other than for group randomization. Surgical management of patients in the hospitals will also be standardized. Postoperative parameters will include pain intensity, rescue analgesic (morphine) consumption, surgical complications (e.g., re-operation, surgical site infection, or bleeding), other perioperative complications (e.g., deep vein thrombosis, cardiac complications, or chest infections), cancer recurrence diagnosed by CT or MRI (done yearly over 5 years) and mortality, both cancer-related and all-cause mortality. In addition, blood will be taken preoperatively for analysis of the following inflammatory and immunological markers:

VEGF will be determined in peritoneal fluid and in serum during surgery. HIF-1A will be determined by immunohistochemistry and microRNA measurements in normal and neoplastic colonic mucosa.

In addition, the microRNA mi21 will be analyzed in by quantitative reverse transcriptase-PCR in colon adenocarcinomas and adjacent non-cancerous tissues.

The CTC in whole blood (in 5-7.5 ml) will be measured with the CellSearch System, according to the manufacturer´s instructions, and the Cell Tracks Analyzer II (Cristofanilli M et al. N Engl J Med 2004:351:781-91).

Inflammatory mediator assay-ELISA Patient serum or EDTA/Heparin plasma will be assessed for cytokine levels by a Luminex multiplex assay (Human Inflammation 12-Plex kit; GM.CSF, IFN-g, IL-1b, IL-2, IL-4, IL-5, IL-6, IL-8, IL-10, IL-12, TNF-a and VEGF from R&D system) and PGE2 levels will be measured by an ELISA kit from Cayman Chemicals Company. In addition, markers of systemic inflammatory response, including CRP, white blood cell count, differential count and total platelet count, will also be measured before and after surgery.

ELIGIBILITY:
Inclusion Criteria:

* ASA status 1-3
* Age group 40-80 years old
* Undergoing elective surgery for colorectal cancer

Exclusion Criteria:

* All contraindications to epidural analgesia
* Chronic opiate medication/drug abuse
* Allergy to morphine

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 221 (Actual)
Dates: Start 2011-03; Primary Completion 2020-12 (Actual); Study Completion 2021-01 (Actual)

PRIMARY OUTCOMES:
Long-term (up to 5 yrs) all-cause mortality | 7 years from start of enrollment
  Cancer specific as well as all-cause mortality would be recorded.

SECONDARY OUTCOMES:
Cancer recurrence detected by MRI; perioperative complications | 7 years following start of enrollment
  All complications during the perioperative period including cancer recurrence detected by MRI examination once each year would be recorded.

OTHER OUTCOMES:
Inflammation | 0-5 days
  Perioperative cytokine concentration in blood assessed between randomised groups as well as surgical technique after 100 recruited patients
Postoperative pain and early recovery | 0 - 7 days postoperatively
  Aspects of early postoperative recovery until discharge would be measured after 200 recruited patients between randomised groups as well as surgical techniques

CONTACTS AND LOCATIONS:
Locations (2):
- Sweden (2):
  - University Hospital, Linköping
  - University Hospital, Örebro